CLINICAL TRIAL: NCT04707989
Title: A Randomized, Placebo Controlled, Study to Evaluate the Tolerance and Safety of a Ketone- Promoting Food Ingredient in Healthy Men and Women
Brief Title: Tolerance and Safety of a Ketone-Promoting Food Ingredient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BHB Therapeutics, Ireland LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KEET-2; BIO-2103 (Other: Biofortis)
Record Dates: First submitted 2020-12-29; First posted 2021-01-13 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Tolerance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone-Promoting Food Ingredient 1 (Experimental): Novel ketone-promoting food ingredient (#1) administered in a beverage once daily for 28 days.
  Interventions: Other: Ketone- Promoting Food Ingredient #1
- Ketone Free Placebo (Placebo Comparator): Beverage matched for appearance, volume, taste and texture to experimental arm (ketone promoting food ingredient #1) that does NOT contain a ketone ingredient. Consumed once daily for 28 days.
  Interventions: Other: Ketone Free Placebo
- Ketone-Promoting Food Ingredient 2 (Active Comparator): Previously characterized ketone-promoting food ingredient (#2) administered in a beverage once daily for 28 days.
  Interventions: Other: Ketone- Promoting Food Ingredient #2

INTERVENTIONS:
Other: Ketone- Promoting Food Ingredient #1 — Novel proprietary food ingredient (#1) that contains precursors to naturally occurring energy molecules called ketone bodies. Promotes mildly elevated blood ketone concentrations. Mixed into a beverage.
  Arms: Ketone-Promoting Food Ingredient 1
Other: Ketone- Promoting Food Ingredient #2 — Previously characterized proprietary food ingredient (#2) that contains precursors to naturally occurring energy molecules called ketone bodies. Promotes mildly elevated blood ketone concentrations. Mixed into a beverage.
  Arms: Ketone-Promoting Food Ingredient 2
Other: Ketone Free Placebo — Beverage that is matched to ketone-promoting food ingredient #1 beverage for appearance, taste, texture and volume. Does not contain ketones or ketone precursors.
  Arms: Ketone Free Placebo

SUMMARY:
The objective of this study is to capture information on tolerance and safety of a ketone-promoting food ingredient in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is generally healthy male or female, 18-65 years of age.
2. Subject has a BMI 18.5-34.9 kg/m2 (inclusive).
3. Subject is willing and able to comply with all study procedures including consumption of breakfast and lunch daily, maintenance of habitual dietary intake, exercise and medication and supplement use, blood draws and the following prior to test visits: fasting (>10 h; water only), no alcohol (>10 h), no cannabis products (>10 h) and no exercise (>10 h).
4. Subject has internet access via computer, phone, or other device and is able to maintain internet access throughout the trial in order to complete online daily questionnaires.
5. Subject has no health conditions that would prevent him from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
6. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject has an abnormal laboratory test result(s) of clinical importance at screening, at the discretion of the Clinical Investigator.
2. Subject has a history or presence of uncontrolled and/or clinically important pulmonary, cardiac, hepatic, renal, endocrine (including type 1 and 2 diabetes), hematologic, immunologic, neurologic, psychiatric or biliary disorders at the discretion of the Investigator.
3. Subject has a clinically important gastrointestinal (GI) condition that would potentially interfere with the evaluation of the study beverage.
4. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
5. Subject is a current user of tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 6 months of screening at the equivalent of >5 cigarettes per day.
6. Subject has a history of or strong potential for alcohol or substance abuse.
7. Subject is consistently using prescriptive or over-the counter medications where alcohol is a contraindication at the discretion of the Investigator.
8. Subject has a known allergy, intolerance, or sensitivity to any of the ingredients in the study beverages.
9. Subject has uncontrolled hypertension as defined by the blood pressure measured at screening.
10. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
11. Subject has experienced any major trauma or any other surgical event within three months of screening.
12. Subject has recently used antibiotics.
13. Subject has extreme dietary habits or has used weight-loss medications or programs within 30 days of screening.
14. Subject has used medications known to influence gastrointestinal function within 30 days of screening.
15. Subject consistently uses anti-inflammatory medications (>5 times/week) within 30 days of screening.
16. Subject has used ketone supplements within 30 days of screening.
17. Subject has unstable use of thyroid, antihypertensive, antidepressant, or statin medications within 6 months of screening.
18. Individual has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.
19. Subject works nights or shifts that means it is not possible to maintain a consistent meal schedule during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Long-term tolerance of ketone promoting food ingredient #1 | Day From baseline to Day 28
  Difference between experimental arm (ketone promoting food ingredient #1) vs placebo in composite score of tolerance, assessed by twice daily tolerance questionnaires completed at home.
  Subjects complete a tolerance questionnaire twice daily, to assess the presence of 10 symptoms before and 4-6h after consuming the study beverage. Questionnaire ranks severity (None, mild, moderate, severe) and incidence (usually, somewhat more than usual, much more than usual). Answers are assigned a numerical value, where higher score is a greater severity and incidence of symptoms. The difference is calculated between the pre- and post- beverage questionnaire for a daily score. Daily scores for the duration of the study are added together to give a single composite score for the whole study period.

SECONDARY OUTCOMES:
Acute tolerance of ketone promoting food ingredient #1 | Days 0, 7 and 14
  Difference between experimental arm (ketone promoting food ingredient #1) vs placebo in composite scores of tolerability, assessed by a tolerance questionnaire at 1h after beverage consumption at clinic visits.
  Subjects complete a tolerance questionnaire twice, to assess the presence of 10 symptoms before and 1h after consuming the study beverage. Questionnaire ranks severity (None, mild, moderate, severe) and incidence (usually, somewhat more than usual, much more than usual). Answers are assigned a numerical value, where higher score is a greater severity and incidence of symptoms. The difference is calculated between the pre- and post- beverage questionnaire for a score representing acute tolerance.
Subjective Arousal after ketone promoting food ingredient #1 | From baseline to Day 28
  Difference between experimental arm (ketone promoting food ingredient #1) vs placebo in the composite scores of the stimulatory and sedative subscale using the Brief Biphasic Alcohol Effect Scale (B-BAES); completed twice daily at home.
  B-BAES presents 6 items in alphabetical order, and subjects rank them on an 11 point scale, from 0 = not at all to 10 = extremely.
  The difference is calculated between the pre- and post- beverage questionnaire for a daily score. Daily scores for the duration of the study are added together to give a single composite score for the whole study period.
  Rueger, S. Y. and A. C. King (2013). "Validation of the brief Biphasic Alcohol Effects Scale (B-BAES)." Alcohol Clin Exp Res 37(3): 470-476.
Safety Blood Profile | From baseline to Day 28
  Change from baseline Day 28 in the incidence of abnormal laboratory test results

OTHER OUTCOMES:
Long-term tolerance of ketone promoting food ingredient #2 | From baseline to Day 28
  Difference between active comparator arm (ketone promoting food ingredient #2) vs placebo in composite score of tolerance, assessed by twice daily tolerance questionnaires completed at home.
  Subjects complete a tolerance questionnaire twice daily, to assess the presence of 10 symptoms before and 4-6h after consuming the study beverage. Questionnaire ranks severity (None, mild, moderate, severe) and incidence (usually, somewhat more than usual, much more than usual). Answers are assigned a numerical value, where higher score is a greater severity and incidence of symptoms. The difference is calculated between the pre- and post- beverage questionnaire for a daily score. Daily scores for the duration of the study are added together to give a single composite score for the whole study period.
Acute tolerance of ketone promoting food ingredient #2 | Days 0, 7 and 14
  Difference between active comparator arm (ketone promoting food ingredient #2) vs placebo in composite scores of tolerability, assessed by a tolerance questionnaire at 1h after beverage consumption at clinic visits.
  Subjects complete a tolerance questionnaire twice, to assess the presence of 10 symptoms before and 1h after consuming the study beverage. Questionnaire ranks severity (None, mild, moderate, severe) and incidence (usually, somewhat more than usual, much more than usual). Answers are assigned a numerical value, where higher score is a greater severity and incidence of symptoms. The difference is calculated between the pre- and post- beverage questionnaire for a score representing acute tolerance.
Subjective Arousal after ketone promoting food ingredient #2 | From baseline to Day 28
  Difference between active comparator arm (ketone promoting food ingredient #2) vs placebo in the composite scores of the stimulatory and sedative subscale using the Brief Biphasic Alcohol Effect Scale (B-BAES); completed twice daily at home.
  B-BAES presents 6 items in alphabetical order, and subjects rank them on an 11 point scale, from 0 = not at all to 10 = extremely.
  The difference is calculated between the pre- and post- beverage questionnaire for a daily score. Daily scores for the duration of the study are added together to give a single composite score for the whole study period.
  Rueger, S. Y. and A. C. King (2013). "Validation of the brief Biphasic Alcohol Effects Scale (B-BAES)." Alcohol Clin Exp Res 37(3): 470-476.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rueger SY, King AC. Validation of the brief Biphasic Alcohol Effects Scale (B-BAES). Alcohol Clin Exp Res. 2013 Mar;37(3):470-6. doi: 10.1111/j.1530-0277.2012.01941.x. Epub 2012 Oct 18. PMID 23078583